CLINICAL TRIAL: NCT05361031
Title: Single Center, Open Label, Repeat Intramuscular Administration, 270 Days, Phase I/2a Clinical Trial to Evaluate Safety, Tolerability of Investigational Product (Engensis: VM202) With Charcot-Marie-Tooth Disease Subtype 1A (CMT1A)
Brief Title: The Safety and Tolerability of Engensis (VM202) in Patients With Charcot-Marie-Tooth Disease Subtype 1A (CMT1A)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Helixmith Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VMCMT-001
Record Dates: First submitted 2022-03-31; First posted 2022-05-04 (Actual); Results first posted 2025-05-29 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-08

CONDITIONS: CMT

STUDY DESIGN:
Intervention Model Description: Single center, repeat dose, open label, phase I/IIA clinical study
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Engensis (VM202) (Experimental): 56 (ea) 0.25mg (0.5 mL) injections in each of the left and right lower limbs on Days 0, 14, 90, and 104.
  Interventions: Biological: Engensis (VM202)

INTERVENTIONS:
Biological: Engensis (VM202) — Intramuscular injections

SUMMARY:
To assess the safety and tolerability of the investigational product Engensis (VM202) injected in the weakened lower limb muscles of CMT1A patients

DETAILED DESCRIPTION:
There are no therapeutic agents for CMT to date. Attempts were made to develop therapeutic agents, but efficacy could not be demonstrated in clinical studies. Most of the attempted developments for therapeutic agents targeted alleviating the symptoms of CMT1A by regulating the expression of PMP22. This study will use Engensis (VM202), which is a DNA plasmid that contains novel genomic cDNA hybrid human HGF coding sequence (HGF-X7) expressing two isoforms of HGF, HGF 728 and HGF 723. HGF has been thought of as an angiogenic factor, but it has been recently identified as serving the role of a neurotrophic factor. Moreover, it has been reported that it can contribute to muscle tissue regeneration by targeting on muscles. Considering the pathologic mechanism of CMT, the biological activity of HGF helps peripheral nerve regeneration, relieves muscle atrophy, and reduces pain, so it is highly likely to show a therapeutic effect for CMT.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females ≥ 19 years of age and ≤ 65 years of age
2. Patients with confirmed diagnosis of CMT1A by genetic testing
3. Patients with mild to moderate severity assessed by Charcot Marie Tooth Neuropathy Score version 2 (CMTNS v2) with a score > 2 and ≤ 20
4. Individuals with lower limb muscle weakness with minimum dorsiflexion or more
5. Individuals who voluntarily consented to participate in this study and signed the IRB approved informed consent form after listening to a description on the characteristics of this clinical study prior to all screening tests
6. Individuals who can comply with the requirements in the clinical study
7. In case of females of child bearing potential, those who test negative in a urine or serum pregnancy test at screening
8. Individuals who practice medically approved contraceptive methods throughout the clinical study

Exclusion Criteria:

1. Patients with significant respiratory, circulatory, renal, gastrointestinal, hepatic, endocrine, hematologic, psychiatric disorders or other severe diseases, or alcohol or drug addiction who may develop safety issues or cause confusion in the interpretation of the clinical study results as determined by the principal investigator
2. Patients with other neuromuscular diseases or neuropathy-inducing factors: Patients with chronic alcohol addiction, undergoing anticancer chemotherapy, or taking neurotoxic drugs
3. Patients diagnosed with diabetes
4. Patients diagnosed with inflammatory bowel disease
5. Patients with a history of stroke or cerebral ischemic attack within 12 months prior to the screening date
6. Patients with a history of coronary artery disease, such as myocardial infarction and unstable angina pectoris, within 12 months prior to the screening date
7. Morbidly obese patients with body mass index (BMI) ≥ 37
8. Patients who underwent orthopedic surgery (corrective surgery for bone and ligament, artificial joint implantation, osteosynthesis, osteotomy, arthroscopic surgery) in the lower limbs within 6 months prior to the screening date
9. Patients who may be affected by the muscle strength measurement test due to ankle contracture or surgery
10. Patients with uncontrolled hypertension (if systolic blood pressure is ≥ 160 mmHg or diastolic blood pressure is ≥ 100 mmHg at screening)
11. Patients or patient's immediate family members (parents, siblings, offspring) with a history of malignant tumors within the last 5 years prior to the screening date, excluding basal cell carcinoma or squamous cell carcinoma that occurs on the skin (if it is determined that there is no possibility of relapse after resection), or with a family history of familial adenomatous polyposis (FAP) or hereditary nonpolyposis colorectal cancer (HNPCC)
12. Patients who have not completed a national cancer screening program applicable to their sex and age (if it cannot be confirmed that the relevant test was received at a national cancer screening center or a recognized screening center)

    However, if it is confirmed that the relevant test was received at a national cancer screening center or a recognized screening center during the screening period, and that the results were within normal range, the patients may participate in the clinical study.

    Common to males and females: If a patient is ≥ 50 years of age, the results of a colonoscopy within 5 years prior to the screening must be determined as being within normal range, and if adenomatous polyps are evident, the results of a colonoscopy within 1 year must be determined as being within normal range (inflammatory polyps or hyperplastic polyps are included in the normal range). If a patient is ≥ 40 years of age, the results of a gastroscopy within 2 years prior to the screening must be within normal range. If a patient is ≥ 54 years of age and has a 30 pack-year history of smoking or more, the results of a low-dose chest CT within 2 years prior to the screening must be within normal range. In case of liver cancer, carriers of hepatitis B or hepatitis C virus and patients with hepatic cirrhosis fall under the exclusion criteria.

    Females: For females ≥ 40 years of age, normal range findings must be confirmed in a mammogram within 2 years. For females ≥ 20 years of age, normal range findings must be confirmed in a Pap smear within 2 years.
13. Patients diagnosed with active pulmonary tuberculosis
14. Patients with HBV or HCV
15. Patients who test positive in human immunodeficiency virus (HIV) antibody test
16. Patients in an immunosuppressive state due to treatments such as immunosuppressants, chemotherapy, and radiotherapy
17. Patients with a history of mental disease within 6 months prior to the screening date, which may interfere with participation in the study
18. Patients who must take medications, that are known to have significant drug interactions within 14 days after the first administration of the investigational product or deemed unsuitable by the investigator's judgment
19. Individuals who participated in another clinical study within 6 months before the time of screening
20. Individuals who have shown significant adverse events such as hypersensitivity reactions to the investigational product
21. Pregnant or breastfeeding females
22. Other individuals determined ineligible by the principal investigator to participate in the clinical study due to other reasons including clinical laboratory test results

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2022-02-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Engensis (VM202)
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Engensis (VM202)
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 40.17 (14.81)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  South Korea | 12

OUTCOME MEASURES:

1. Primary Outcome: Safety of Intramuscular (IM) Injections of Engensis in Participants
Description: Frequency and percentage of treatment-emergent adverse events (TEAEs) and serious adverse events after injections, injection site reactions, vital sign, and clinically significant laboratory values for Engensis.
Time Frame: Day 0 visit to the Day 270 visit
Population: Safety population
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis (VM202)
Number analyzed (Participants) | 12
Participants
  Injection site pruritis | 1
  Oedema peripheral | 1
  Pneumonia | 1
  Uterine leiomyoma | 1

2. Secondary Outcome: Evaluation of Severity of Disease Changes Following Engensis Injections - Charcot Marie Tooth Neuropathy Score Version 2
Description: Charcot-Marie-Tooth Neuropathy Score version 2 is a measurement tool for evaluating the severity of disease. The scoring system is the total neuropathy score, by assessing the symptoms of Charcot-Marie-Tooth patients due to sensory impairment. Measurements were performed in three items for the symptoms of disease, four items for the signs, and two items for neurophysiological testing, a total of nine separate test items.
  The Total Severity Score is the summed scores of all subscores and has a total minimum score of 0 and a maximum score of 36. The Total Severity Score Scale of the disease is classified according to the Total Score as either mild (0 to 10), moderate (11 to 20), or severe (20 to 36).
  The Change from Baseline Total Severity Score is the difference between the Day 0 and the Day 270 scores.
  A negative difference in the Total Severity Score Change from Baseline to Day 270, indicates an improvement of the treated groups' total severity level.
Time Frame: Day 0 and Day 270
Population: Total Severity Score, and Change from Baseline of Total Severity Score of disease: Charcot-Marie-Tooth Neuropathy Score-version 2 - Intent to Treat population from Day 0 to Day 270.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Engensis (VM202): 56 (ea) 0.25mg (0.5 mL) injections in each of the left and right lower limbs on Days 0 and Day 270.
  Engensis (VM202): Intramuscular injections
Arm/Group | Engensis (VM202)
Number analyzed (Participants) | 12
score on a scale
  Day 0 - Total Severity Score | 15.58 (3.37)
  Day 270 - Total Severity Score | 13.42 (2.75)
  Day 270 - Change from Baseline of Total Severity Scores | -2.17 (1.11)

3. Secondary Outcome: Evaluation of Patient's Neurological Disability - Functional Disability Score
Description: Change from Baseline (Day 0) in Functional Disability Scale at Days 90, 180, and 270; as assessed using the Functional Disability Scale 0 - 8 points, where normal is 0 point, best case, and if determined as bedridden, it is evaluated as 8 points, worst case.
  0=normal; 1=cramps and fatigability; 2=inability to run; 3=possible unaided; 4=with cane; 5=with crutch; 6=with walker; 7=wheelchair; 8=bedridden.
  Changes in severity of disease: Functional Disability Scale - Intent-to-Treat population.
Time Frame: Day 0, 90, 180 and Day 270
Population: Changes in severity of disease: Functional Disability Scale - Intent-to-Treat population
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Engensis (VM202)
Number analyzed (Participants) | 12
score on a scale
  Day 90 | 0.08 (0.29)
  Day 180 | -0.25 (0.45)
  Day 270 | -0.58 (0.51)

4. Secondary Outcome: Evaluation of the Activity Level of Patients With Peripheral Neuropathy Using the Overall Neuropathy Limitation Score Leg Scale
Description: Change from baseline (Day 0) in the overall neuropathy limitation score leg scale at Days 90, 180, and 270. The Overall Neuropathy Limitation Score is scored from 0 to 7. The worst score, 7 points, is defined as restricted to wheelchair, or bed most of the day, unable to make any purposeful movements of the leg.
Time Frame: Day 0, 90, 180 and Day 270
Population: Intent to Treat population
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Engensis (VM202)
Number analyzed (Participants) | 12
units on a scale
  Day 90 | -0.08 (0.29)
  Day 180 | -0.08 (0.29)
  Day 270 | -0.33 (0.49)

5. Secondary Outcome: Evaluation of Patient's Walking Ability - Change From Baseline in the 10-Meter Walk Test
Description: This test measures the time in seconds required for a subject to walk 10 meters through the 10-Meter Walking Test version 2.2.
  Changes in the Mean Time in seconds for lower limb function assessment: 10 Meter Walk Test - Intent to Treat population, from Day 0 to Days 90, 180, and 270. The larger the change in time (Seconds) from Day 0 to Visit date indicates a worsening of the patients walking ability.
Time Frame: Day 0, 90, 180 and Day 270
Population: Changes in the mean time in seconds for lower limb function assessment: 10 Meter Walk Test - Intent to Treat population, from Day 0 to Days 90, 180, and 270
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Engensis (VM202)
Number analyzed (Participants) | 12
Seconds
  Day 90 | 0.02 (0.15)
  Day 180 | 0.08 (0.20)
  Day 270 | 0.06 (0.20)

6. Secondary Outcome: Changes in Fatty Infiltration Level of Lower Limb Muscles
Description: Changes from baseline (Day 0) in the fat content of lower limb muscles at Day 270.
  The muscles of lower limbs were imaged with Magnetic Resonance Imaging leg scan, and the degree of fatty infiltration of the leg muscles injected with the investigational product was measured and valuated as fat content value (percent) at one level for each muscle. The six MRI imaging sites to be measured were as follows: peroneus longus left/right, gastrocnemius left/right, and tibialis anterior left/right.
Time Frame: Day 0 and Day 270
Population: Intent to Treat population
Measure: Mean (Standard Deviation); unit: percentage fat content
Arm/Group | Engensis (VM202)
Number analyzed (Participants) | 12
percentage fat content
  Right peroneus longus | 1.79 (3.36)
  Right gastrocnemius | 0.22 (1.66)
  Right tibialis anterior | 1.91 (2.34)
  Left peroneus longus | 3.21 (6.66)
  Left gastrocnemius | 0.24 (2.53)
  Left tibialis anterior | 0.07 (2.83)

7. Secondary Outcome: Change From Baseline in Nerve Conduction Velocity at Day 270
Description: Change from baseline in Nerve Conduction Velocity to Day 270, for evaluation of the presence of a disorder in a neurotransmission pathway, as assessed using the Nerve Conduction Study version 2.0
  Nerve regeneration potential (Electroneurography): Nerve Conduction Velocity (measured in meters per second) - Intent-to-Treat population. Larger negative change from baseline values indicates a slowing of the Nerve Conduction Velocity which is a worsening of the electroconduction function of the specified nerve.
Time Frame: Day 0 and Day 270
Population: Intent-to-Treat population
Measure: Mean (Standard Deviation); unit: meters/second
Arm/Group | Engensis (VM202)
Number analyzed (Participants) | 12
meters/second
  Right median nerve | 0.08 (1.73)
  Right ulnar nerve | 0 (2.04)
  Right radial nerve | -1.25 (2.90)
  Right tibial nerve | -0.25 (1.86)
  Right peroneal nerve | 1.33 (4.31)
  Right sural nerve | -0.17 (0.39)
  Left median nerve | 0.25 (1.36)
  Left ulnar nerve | -0.08 (1.83)
  Left radial nerve | -1.83 (5.54)
  Left tibial nerve | 1.33 (6.21)
  Left peroneal nerve | -1.33 (4.44)
  Left sural nerve | -0.33 (0.78)

8. Secondary Outcome: Numbers of Participants With and Without Hepatocyte Growth Factor Antibody Generation in the Body at Baseline (Day 0) and Day 270.
Description: The presence of hepatocyte growth factor antibody generation by Engensis (VM202) assessed using anti-hepatocyte growth factor antibody test at Day 0 and Day 270
Time Frame: Day 0 and Day 270
Population: Intent to Treat population
Measure: Count of Participants; unit: Participants
Arm/Group | Engensis (VM202)
Number analyzed (Participants) | 12
Participants
  Yes - HGF antibody present at baseline | 0
  Yes - presence of HGF antibody at Day 270 | 0
  No - HGF antibody not present at baseline | 12
  No - HGF antibody not present at Day 270 | 12

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from the Day 0 visit to the Day 270 visit
Arm/Group | Engensis (VM202)
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 3/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engensis (VM202) (N=12)
pneumonia (Infections and infestations) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Engensis (VM202) (N=12)
Injection site pruritis (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
pneumonia (Infections and infestations) | 1 (1)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-06-07): https://cdn.clinicaltrials.gov/large-docs/31/NCT05361031/Prot_000.pdf
  • Statistical Analysis Plan (2021-10-18): https://cdn.clinicaltrials.gov/large-docs/31/NCT05361031/SAP_001.pdf